CLINICAL TRIAL: NCT01310088
Title: Blood Pressure and Central Vascular Stiffness in Obese Children. Relationship to Metabolic Disturbances and Subclinical Cardiovascular Damage. Effect of Weight Reduction
Acronym: AORTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Kristian Hvidt / MD, Division of Cardiology, Department of Medicine, Holbaek Hospital, University of Copenhagen, Denmark
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AORTA-SJ-166
Record Dates: First submitted 2011-02-28; First posted 2011-03-07 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Central Blood Pressure; Obesity; Subclinical Organ Damage; Children; Adolescent
Keywords: Childhood; Child; adolescent; central blood pressure; ambulatory blood pressure monitoring; ABPM; clinic blood pressure; pulse wave velocity; PWV; Pulse cave analysis; PWA; heart rate variability; HRV; Echocardiography; Urine microalbuminuria; blood samples
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Experimental): Treatment protocol The Children's Obesity Clinic Department of Paediatrics Holbaek Hospital, University of Copenhagen Denmark
  Interventions: Behavioral: Lifestyle intervention
- Control (No Intervention): Healthy age and gender matched control subjects. Recruited from school visits.

INTERVENTIONS:
Behavioral: Lifestyle intervention — Treatment protocol. The Children's Obesity Clinic Department of Paediatrics Holbaek Hospital, University of Copenhagen Denmark
  Arms: Lifestyle counseling

SUMMARY:
The global epidemic of obesity in childhood continues to evolve and threaten future health and life expectancy primarily due to the increased incidence of cardiovascular disease. Obesity is strongly related to high blood pressure (hypertension) and both conditions pose a risk for target organ damage, which can follow a subject from childhood into adult life. The AORTA study will investigate central hemodynamics and organ damage in 100 obese children and adolescents in order to gain insight to the complex interplay of hypertension, obesity and subclinical damage in order to intensify more precise prevention, thereby reducing the future development of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* age 10-18
* BMI for age and sex above 95 percentile
* referred for treatment at the The Children's Obesity Clinic, Department of Paediatrics, Holbaek Hospital, University of Copenhagen
* oral and written consent by their parents

Exclusion Criteria:

* children who can not cooperate to DEXA scanning or other procedures
* linguistic difficulties that impair communication

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Central Blood Pressure | one year follow up
  Obtained by the SphygmoCor Device, software version 9, AtCor Medical, Australia.

SECONDARY OUTCOMES:
Pulse Wave velocity | one year follow up
  Measured in meters per second.
Ambulatory Blood Pressure Monitoring and Clinic Blood Pressure | one year follow up
  Measured in milimeters of mercury (mm Hg). Analysed into Blood Pressure standard deviation scores (BP SDS).
  Ambulatory Blood Pressure Monitoring (ABPM) is analysed into Amulatory Arterial Stiffness Index (AASI). ASSI is 1 minus the correlation coefficient when the Systolic Blood Pressure is plottet agiant the diastolic Blood Pressure from a ABPM.
Heart Rate variability | one year follow up
Metabolic and Cardiovascular Blood Samples | one year follow up
Urine Albumine-Creatinine Ratio (UACR) | one year follow up
  Microalbuminuria (MAU) defined by urine albumine-creatinine ratio (UACR) ≥ 3,5 mg/mmol (women) and 2,5 mg/mmol (men). Mean of two morning spot urine samples.
Echocardiography and ultrasound of aortic wall distensibility | one year follow up
Electrocardiography | one year follow up
  Conventional 12 lead electrocardiography (ECG). Analysis of:
  * Heart rate (beats per minute)
  * P waves, QRS waves, ST segment and T waves (durations: miliseconds, amplitude: milimeters/Voltage)
  * Intervals: PQ, PR, QRS, ST, T waves (miliseconds)
  * Configuration of the T wave.
Dual energy X-ray absorptionmetry (DEXA scan) | one year follow up
  A full body DEXA scan gives precise knowlegde of the body fat mass and fat free mass. Fat mass can be converted into fat mass index and fat free mass can be converted into fat free mass index, besides BMI standard deviation score (BMI SDS).
  A DEXA scan also gives information on bone mineral density (BMD), a parameter of bone status, and regional estimates: truncus, abdomen, thorax, arms and legs.
Anthropometric measures | one year follow up
  Height, Waist, Weight, BMI (weight/height²)

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Hvidt, MD, Principal Investigator — Division of Cardiology, Department of Medicine, Holbaek Hospital, University of Copenhagen, Denmark; Hans Ibsen, DMSc, MD, Study Chair — Division of Cardiology, Department of Medicine, Holbaek Hospital, University of Copenhagen; Jens-Christian Holm, PhD, MD, Study Director — The Children's Obesity Clinic, Department of Paediatrics, Holbaek Hospital, University of Copenhagen; Michael Hecht Olsen, DMSc, PhD, MD, Study Director — Division of Cardiology, Department of Medicine, Glostrup Hospital, University of Copenhagen
Locations (2):
- Denmark (2):
  - Division of Cardiology, Department of Medicine, Holbaek Hospital, University of Copenhagen, Holbæk
  - The Children's Obesity Clinic, Department of Paediatrics, Holbaek Hospital, University of Copenhagen, Holbæk

REFERENCES:
- [Background] Han JC, Lawlor DA, Kimm SY. Childhood obesity. Lancet. 2010 May 15;375(9727):1737-48. doi: 10.1016/S0140-6736(10)60171-7. Epub 2010 May 5. PMID 20451244
- [Background] Singh AS, Mulder C, Twisk JW, van Mechelen W, Chinapaw MJ. Tracking of childhood overweight into adulthood: a systematic review of the literature. Obes Rev. 2008 Sep;9(5):474-88. doi: 10.1111/j.1467-789X.2008.00475.x. Epub 2008 Mar 5. PMID 18331423
- [Background] Stabouli S, Kotsis V, Zakopoulos N. Ambulatory blood pressure monitoring and target organ damage in pediatrics. J Hypertens. 2007 Oct;25(10):1979-86. doi: 10.1097/HJH.0b013e3282775992. PMID 17885534
- [Background] Hansen TW, Jeppesen J, Rasmussen S, Ibsen H, Torp-Pedersen C. Ambulatory blood pressure monitoring and risk of cardiovascular disease: a population based study. Am J Hypertens. 2006 Mar;19(3):243-50. doi: 10.1016/j.amjhyper.2005.09.018. PMID 16500508
- [Background] Litwin M, Niemirska A, Ruzicka M, Feber J. White coat hypertension in children: not rare and not benign? J Am Soc Hypertens. 2009 Nov-Dec;3(6):416-23. doi: 10.1016/j.jash.2009.10.002. PMID 20409984
- [Background] Hansen TW, Jeppesen J, Rasmussen S, Ibsen H, Torp-Pedersen C. Relation between insulin and aortic stiffness: a population-based study. J Hum Hypertens. 2004 Jan;18(1):1-7. doi: 10.1038/sj.jhh.1001620. PMID 14688804
- [Background] Willum-Hansen T, Staessen JA, Torp-Pedersen C, Rasmussen S, Thijs L, Ibsen H, Jeppesen J. Prognostic value of aortic pulse wave velocity as index of arterial stiffness in the general population. Circulation. 2006 Feb 7;113(5):664-70. doi: 10.1161/CIRCULATIONAHA.105.579342. PMID 16461839
- [Background] Vitarelli A, Giordano M, Germano G, Pergolini M, Cicconetti P, Tomei F, Sancini A, Battaglia D, Dettori O, Capotosto L, De Cicco V, De Maio M, Vitarelli M, Bruno P. Assessment of ascending aorta wall stiffness in hypertensive patients by tissue Doppler imaging and strain Doppler echocardiography. Heart. 2010 Sep;96(18):1469-74. doi: 10.1136/hrt.2010.198358. Epub 2010 Jul 18. PMID 20643663
- [Derived] Muhamed PK, Olsen MH, Holm JC, Ibsen H, Hvidt KN. Cuff size influences blood pressure measurement in obese children and adolescents. Dan Med J. 2016 Jan;63(1):A5183. PMID 26726900
- [Derived] Hvidt KN, Olsen MH, Holm JC, Ibsen H. Obese children and adolescents have elevated nighttime blood pressure independent of insulin resistance and arterial stiffness. Am J Hypertens. 2014 Nov;27(11):1408-15. doi: 10.1093/ajh/hpu055. Epub 2014 Apr 9. PMID 24717420